CLINICAL TRIAL: NCT07308834
Title: Phase 1/2a Study to Evaluate the Safety and Tolerability Intra-articular CX-011 to Treat Moderate to Severe Pain From Knee Osteoarthritis
Brief Title: Evaluation of Intra-articular CX-011 to Treat Moderate to Severe Pain From Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CarthroniX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX011-2024-001
Record Dates: First submitted 2025-12-22; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis of the Knees
Keywords: OA; Knee; injectable

STUDY DESIGN:
Intervention Model Description: This is a one-center, prospective, randomized, double-blind, placebo-controlled, escalating three dose, Phase 1/2a study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: CX-011
- CX-011 low dose (Experimental)
  Interventions: Drug: CX-011
- CX-011 medium dose (Experimental)
  Interventions: Drug: CX-011
- CX-011 high dose (Experimental)
  Interventions: Drug: CX-011

INTERVENTIONS:
Drug: CX-011 — CX-011 is a hydrophobic small molecule for intra-articular (IA) administration that is being developed for the treatment of subjects with osteoarthritis of the knee.

SUMMARY:
Study is designed to evaluate the safety and effectiveness of a drug called CX-011 to treat pain in patients with osteoarthritis of the knee. Osteoarthritis produces pain in the knee (and other joints) that typically is worsened by activities such as long distance walking and is alleviated by rest.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the safety and tolerability of three escalating doses of CX-011 (100, 300, and 1000 μg) following a single intra-articular administration. Safety assessments will include the incidence and severity of local and systemic adverse events, procedure- and product-related serious adverse events, physical examinations, index knee evaluations, vital signs, electrocardiograms, and safety laboratory tests. Dose-limiting toxicities and the maximum tolerated dose will be determined based on these assessments.

Secondary objectives focus on evaluating the preliminary efficacy of CX-011 for the treatment of knee osteoarthritis pain and function, as well as further characterization of its safety profile. Efficacy endpoints include changes from baseline in pain intensity measured by the Visual Analog Scale (VAS) at 4, 12, and 24 weeks post-injection, as well as percentage improvements in the pain and function subscales of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at the same time points.

Up to 72 patients will participate in this study (in one study center). The expected length of participation in the study is about 28 weeks including the screening period.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent to participate in the study.
2. Males or females 18 years of age or less than 75 years old.
3. Diagnosis OA of the index knee by a combination of clinical and radiographic findings wherein the index knee is self-identified by the patient as the more severe knee and symptoms have persisted for 3 months.
4. Radiographic evidence of OA in the tibiofemoral compartment of the index knee (Kellgren-Lawrence grades II or III) within 6 months prior to Screening or during the Screening period.
5. Index knee pain on most days (greater than 15) over the last month
6. Patients who have failed to adequately respond for at least 6 months within the previous 12 months to at least two osteoarthritis therapies that include least 1 pharmacological treatment such as simple analgesics (e.g., acetaminophen); nonsteroidal anti- inflammatory drugs (NSAIDS) conservative, non-pharmacological therapy; avoidance of activities that cause joint pain; exercise; weight loss; physical therapy; and removal of excess fluid from the knee.
7. VAS Pain score of 40-80 on a 0 - 100 scale to be reconfirmed at time of treatment.
8. Overall index knee pain score of 11 or more in the index knee using the 0 - 20 WOMAC Pain scale.
9. hsCRP greater or equal 2 mg/L
10. Body mass index less than 40 kg/m2
11. If female, must not be pregnant or nursing and willing to refrain from becoming pregnant.
12. Willing to agree not to use illicit drugs during the study, and to have illicit drug testing at screening and at later time points if illicit drug use is suspected during the study.
13. Able to comply with study requirements and complete the full sequence of protocol-related procedures and evaluations, including post-hospitalization, outpatient, and follow-up visits and ability to follow verbal and written instructions.

    Exclusion Criteria:
14. Daily use of assistive devices (e.g. cane or walker) or presence of comorbidities that would limit the patient's ability to walk.
15. History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis or amyloidosis.
16. Unstable joint (such as a torn anterior cruciate ligament)
17. Inability to undergo Magnetic Resonance Imaging (MRI) due to presence of surgical hardware or other foreign body in the index knee, or because of patient's claustrophobia
18. Regular use of anticoagulants
19. Symptoms of locking, intermittent block to range of motion, or loose body sensation that could indicate meniscal displacement or an IA loose body; knee ligament instability.
20. Major dysplasias or congenital abnormalities
21. Corticosteroid injection into the index knee within 3 months prior to screening; extended-release steroid use within 4 months prior to screening.
22. Viscosupplement (e.g., hyaluronic acid [HA]) injection, platelet-rich plasma injection, bone marrow aspirate or bone marrow aspiration concentrate, placental-derived tissue/cells, adipose tissue, or any other autologous or allogeneic product) into the index knee within 3 months prior to screening.
23. Knee surgery or procedure on the index knee within 12 months prior to screening and/or planned knee surgery during the study including cold or radiofrequency nerve ablation.
24. Knee surgery or procedure on the contralateral knee within 6 months prior to screening and/or planned knee surgery during the study including cold or radiofrequency nerve ablation.
25. Acute index knee trauma within 3 months prior to screening.
26. Knee joint infections, skin diseases or infections in the area of the injection site.
27. Current therapy with any immunosuppressive therapy, including corticosteroids (> 5 mg/day of prednisone) or patients with conditions that would likely include treatment with immunosuppressive therapy (including corticosteroids) during the study period.
28. HbA1c > 8% and/or insulin-dependent diabetes
29. Average systolic BP > 160 mmHg or diastolic BP > 100 mmHg on > 3 blood pressure medications.
30. Clinically significant findings on physical examination or screening tests (e.g. laboratory and radiographic) that are not specific to OA of the knee and may interfere with study conduct or interpretation of data or increase patient risk.
31. Clinically significant intercurrent illness, medical condition, non-knee pain, or medical history (including neurological or mental illness, human immunodeficiency virus, autoimmune diseases or connective tissue disorder, fibromyalgia, complex regional pain syndrome, clinical anxiety, clinical depression, any active infection including hepatitis B or C) that would jeopardize patient safety, limit participation, or compromise interpretation of data derived from the patient.
32. Participation in another clinical trial within the previous 30 days before screening or planned participation in another clinical trial within the study period

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine tolerability by monitoring the frequency of treatment-emergent adverse events | 24 weeks
  Tolerability will be measured by the incidence and severity of dose-limiting toxicity events as well as the incidence and severity of local and systemic adverse events (AEs)
Composite safety profile of CX-011 based on change from baseline in clinical laboratory parameters | 24 weeks
  The incidence and severity of clinically-significant laboratory findings determined by change from baseline in blood chemistry, hematology and urinalysis as indicators of blood, liver and kidney function, respectively.

SECONDARY OUTCOMES:
Pain (Visual Analog Scale, VAS) | 24 weeks
  Determine the change from baseline to 4, 12 and 24 weeks in the Visual Analog Scale (VAS), with scores ranging from 0-100; lower scores represent better outcomes.
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 24 weeks
  Determine the percent improvement in the Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain and function subscales at 4, 12 and 24 weeks. Scores for the pain subscale range from 0-20, while scores for the function subscale range from 0-68; lower scores reflect better outcomes.

IPD SHARING:
Plan to Share IPD: Undecided
IPD in this study could represent proprietary information; once the study has been completed, the release of IPD will be re-evaluated.